CLINICAL TRIAL: NCT01635556
Title: Evaluation of a Modified Dialectical Behavior Therapy Program for Borderline Personality Disorder
Brief Title: Evaluation of a Modified Dialectical Behavior Therapy Program
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: H2012:128
Record Dates: First submitted 2012-05-23; First posted 2012-07-09 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2014-11

CONDITIONS: Borderline Personality Disorder
Keywords: borderline personality disorder; dialectical behavior therapy; psychological treatment
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Dialectical Behavior therapy — Weekly psychotherapy of both individual and group sessions

SUMMARY:
The goal of this pilot project is to offer outpatient Dialectical Behavior Therapy (DBT) treatment as described in Linehan's text (1993), which is considered an effective treatment of borderline personality disorder. This treatment consists of weekly individual psychotherapy, weekly group skills training, 24 hour telephone consultation, and weekly team consultation meetings for therapists. The investigators program is able to offer all of these components except the 24 hour phone consultation (which has been modified due to employment/union guidelines of interdisciplinary staff working within the investigators health care system). This project intends to offer the treatment for a period of 6 months.

As such, this proposed research project seeks to assess the feasibility of implementing an outpatient DBT program within a public health care setting in Canada. This study also aims to evaluate this DBT program for clinical effectiveness in its modified format. Specifically, the investigators will examine relevant outcomes related to patient functioning (e.g., depression, self-harm and suicidal behaviors, and admissions to hospital/ER visits) and improvement (e.g., improved quality of life, meeting work/employment goals) pre and post completion of this 6 month treatment program.

The investigators hypotheses are that each patient will show improvement in all outcome variables (e.g., improved mood and quality of life, decreased self-harm, decreased ER visits and hospitalization visits, etc). The investigators also hypothesize that the investigators modified program will produce comparable results to those from studies of standard outpatient DBT.

DETAILED DESCRIPTION:
Standard DBT includes four modes of intervention: weekly individual psychotherapy; weekly skills group; 24 hour phone consultation to the patient; and consultation team meetings. The skills group is focused on teaching skills (mindfulness, emotional regulation, distress tolerance, and interpersonal effectiveness), and facilitating the replacement of maladaptive behaviors with adaptive behaviors (Neasciu, Rizvi, & Linehan, 2010). Individual therapy sessions focus on reducing target problem behaviors (e.g., life threatening behavior, therapy interfering behavior, quality of life interfering behaviors). Phone consultation is to aid the client in generalizing skill use to their every day life. The consultation team meetings are for the therapists, to provide support, and to aid therapists in staying adherent to a DBT frame of treatment.

This project will be utilizing a convenience sample. Patients are referred to the program by their psychiatrist/family doctor. They are assessed by a Clinical Psychologist to determine if they meet criteria for a diagnosis of Borderline Personality Disorder via clinical interview and a semi-structured diagnostic interview. They must also meet the inclusion/exclusion criteria for participation in the program, which are as follows:

Inclusion Criteria

* 18 years or older
* Borderline personality disorder diagnosis
* Chronic suicidal ideation or parasuicidal acts, or other self-destructive, impulsive behaviors
* Must be willing to sign DBT contract and commit to 6-month duration of treatment of both individual therapy and skills training group.

Exclusion Criteria

* Active psychosis
* Severe developmental delays, cognitive impairment or learning disabilities
* No violent behaviors will be tolerated. Patients with a history of dangerous or aggressive behaviors towards others, history of medical harm to previous therapists may not be considered.

Following this, they must agree to participate in the program and to the program requirements (weekly individual therapy, skills group, etc). Once this has occurred, they will be approached by a research assistant to discuss with them their voluntary participation in this research study. Once consent is provided, the patient will complete several baseline measures. These same measures will be completed at post treatment (6 months) and then again at 12 months and 18 months for follow-up. Each patient will also complete a weekly diary card, which asks them to record several aspects of daily functioning, as well as self-harm urges and behaviors, and use of skills taught in DBT.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Borderline Personality Disorder
* Chronic suicidal ideation or parasuicidal acts, or other self-destructive, impulsive behaviors
* Must be enrolled in dialectical behavior therapy program

Exclusion Criteria:

* Active psychosis
* Severe developmental delays, cognitive impairment or learning disabilities
* History of or current violent/aggressive behaviors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be selected from the community.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life Enjoyment and Satisfaction Questionnaire | Baseline
  This measure assesses the degree of enjoyment and satisfaction experienced during the past week in several areas: physical health, feelings, work, household duties, school, leisure time, and social relationships.
Quality of Life Enjoyment and Satisfaction Questionnaire | Change - baseline to 6 months
  This measure assesses the degree of enjoyment and satisfaction experienced during the past week in several areas: physical health, feelings, work, household duties, school, leisure time, and social relationships.
Quality of Life Enjoyment and Satisfaction Questionnaire | Change - 6 months to 12 months
  This measure assesses the degree of enjoyment and satisfaction experienced during the past week in several areas: physical health, feelings, work, household duties, school, leisure time, and social relationships.
Quality of Life Enjoyment and Satisfaction Questionnaire | Change - 12 months to 18 months
  This measure assesses the degree of enjoyment and satisfaction experienced during the past week in several areas: physical health, feelings, work, household duties, school, leisure time, and social relationships.

SECONDARY OUTCOMES:
Borderline Symptom List 23 | Baseline
Borderline Symptom List 23 | Change - baseline to 6 months
Borderline Symptom List 23 | Change - 6 months to 12 months
Borderline Symptom List 23 | Chabge - 12 months to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Krysanski, PHD, Principal Investigator — University of Manitoba
Locations (1):
- Victoria General Hospital, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No